CLINICAL TRIAL: NCT05579795
Title: Tethered Cord Syndrome: Surgical Management and Outcome
Brief Title: Surgical Management and Outcome of Tethered Cord Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amr Gamal Hussein Mohamed, Principal Investigator, Assiut University
Other Study IDs: Tethered Cord Syndrome
Record Dates: First submitted 2022-10-03; First posted 2022-10-14 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Tethered Cord Syndrome
MeSH Terms: conditions — Neural Tube Defects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Detethering of the spinal cord — Release of the tethered spinal cord

SUMMARY:
The aim of this study is to assess surgical management and outcome of Tethered cord syndrome

DETAILED DESCRIPTION:
Tethered cord syndrome (TCS) is a developmental abnormality of the neuroaxis which is usually diagnosed in childhood. The actual tethering has been attributed to a variety of pathologic entities, including a thickened tight filum terminale , intradural lipomas with or without a connecting extradural component, intradural fibrous adhesions, diastematomyelia, and adherence of the neural placode following previous closure of a myelomeningocele. However, sufficient differences in the mode of onset, clinical manifestations, and outcome exist between pediatric and adolescent patients with tethered cord to warrant a more detailed analysis of the adult syndrome. The most problematic technical consideration in surgery for the release of the tethered cord is how to preserve functioning neural elements and rebuild the dural sac to avoid CSF leak. The purpose of this study is to review causes of Tethered cord, clinical presentation, diagnostic tools, treatment options and outcome in school-aged children, adolescents, and young adults with Tethered cord.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Tethered cord syndrome presenting at our institute
* Patients with spinal dysraphism
* Lipomyelomeningocele with Tethered cord
* patients presented with neurological deficit after lipomyelomeningocele repair due to Tethered cord
* patients presented with neurological deficit after myelomeningocele repair due to Tethered cord
* Diastematomyelia with Tethered cord - Tethered cord due to filum terminale.
* Tethered cord due to fibrous adhesions

Exclusion Criteria:

* Asymptomatic Patients with Tethered cord discovered accidentally

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Males and Females below 16 years old with Tethered cord syndome
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2022-11-02 (Estimated); Primary Completion 2024-11-02 (Estimated); Study Completion 2024-12-02 (Estimated)

PRIMARY OUTCOMES:
Motor power | Two years
  Outcome of Detethering of the Tethered spinal cord according to Motor power of the lower limbs 5 grades 0: No visible muscle contraction
  1. Visible muscle contraction with no or trace movement
  2. Limb movement, but not against gravity
  3. Movement against gravity but not resistance
  4. Movement against at least some resistance supplied by the examiner
  5. Full strength
Sensations | Two years
  Outcome of Detethering of the Tethered spinal cord according to the sensations of lower limbs , is there decreased sensations of lower limbs and if improved or not
Sphincter's function | Two years
  Outcome of Detethering of the Tethered spinal cord according to is there urinary incontinence or stool incontinence and if improved or not

IPD SHARING:
Plan to Share IPD: Yes
The aim of this study is to assess surgical management and outcome of Tethered cord syndrome.
Supporting Information: CSR
Time Frame: two years